CLINICAL TRIAL: NCT00825500
Title: A Multi-center, Randomized, Double-Blind, Placebo-Controlled, Single Dose Efficacy and Safety Study of Staccato® Loxapine for Inhalation in Outpatients With Migraine Headache
Brief Title: Staccato Loxapine in Migraine (Out Patient)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMDC-104-202; 24-October-2008
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2009-08

CONDITIONS: Migraine Headache
Keywords: Migraine headache; Loxapine; Staccato
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inhaled Placebo (Placebo Comparator): Inhaled Staccato Placebo (0 mg)
  Interventions: Drug: Inhaled Placebo
- Inhaled Loxapine 1.25 mg (Active Comparator): Inhaled Staccato Loxapine 1.25 mg, single dose
  Interventions: Drug: Inhaled Loxapine 1.25 mg
- Inhaled Loxapine 2.5 mg (Experimental): Inhaled Staccato Loxapine 2.5 mg, single dose
  Interventions: Drug: Inhaled Loxapine 2.5 mg

INTERVENTIONS:
Drug: Inhaled Placebo — Inhaled Staccato placebo (0 mg)
  Arms: Inhaled Placebo
Drug: Inhaled Loxapine 1.25 mg — Inhaled Staccato Loxapine 1.25 mg, single dose
  Arms: Inhaled Loxapine 1.25 mg
Drug: Inhaled Loxapine 2.5 mg — Inhaled Staccato Loxapine 1.25 mg, single dose
  Arms: Inhaled Loxapine 2.5 mg

SUMMARY:
Assess the safety and efficacy of Staccato Loxapine in patients with moderate to severe migraine headache with or without aura in an outpatient setting.

DETAILED DESCRIPTION:
This study was designed to compare the safety and pharmacodynamic profiles of concomitant administration of single doses of ADASUVE and intramuscular (IM) lorazepam compared to that of each agent administered alone. Respiratory pharmacodynamics were monitored through recordings of respirations/minute and pulse oximetry. Other pharmacodynamic safety measures included effects on blood pressure, heart rate, sedation, and psychomotor measures of attention, information processing speed, reaction time, and coordination.

ELIGIBILITY:
Inclusion Criteria

* Male or female between the ages of 18 to 65 years, inclusive
* History of migraine headache with or without aura (according to IHS Criteria 1.1 or 1.2 for diagnosis beginning at least 6 months prior to study entry) (International Headache Society Clinical Trials Subcommittee, 2000)
* At least 3 migraine attacks in the last 3 month period (but not more than 8 migraine attacks in the last month)
* Pain rating of moderate or severe (on a none-mild- moderate-severe scale) prior to dosing
* Agreed not to use the study drug within 72 hours of a prior migraine attack
* Agreed not to use any acute migraine or pain medication within 48 hours prior to dosing (including over-the-counter [OTC] products); medications for migraine prophylaxis other than those that were exclusionary were permitted if stable doses had been given for at least 30 days prior to screening
* Agreed not to use medications (including OTC products) for motion sickness, tinnitus, or vertigo within 48 hours prior to dosing.
* Were able to speak, read, and understand English and were willing and able to provide written informed consent on an IRB-approved form prior to the initiation of any study procedures
* Were willing and able to comply with the study schedule and requirements, and agreed to return to the clinic within 5 working days of use of the study drug
* In good general health prior to study participation as determined by a detailed medical history, physical examination, 12-lead electrocardiogram (ECG), blood chemistry profile, hematology, urinalysis, and in the opinion of the investigator
* Female participants (if of child-bearing potential and sexually active) and male participants (if sexually active with a partner of child-bearing potential) who agreed to use a medically acceptable and effective birth control method throughout the study and for 1 week following the end of the study. Medically acceptable methods of contraception that could be used by the participant and/or his/her partner included abstinence, birth control pills or patches, diaphragm with spermicide, intrauterine device (IUD), condom with foam or spermicide, vaginal spermicidal suppository, surgical sterilization, and progestin implant or injection. Prohibited methods included the rhythm method, withdrawal, condoms alone, or diaphragm alone.

Exclusion Criteria

* Use of antipsychotics (including butryophenones, phenothiazines, thioxanthenes, aripiprazle, olanzapine, risperidone), tricyclic antidepressants, trazodone, anticonvulsants (except topiramate), barbiturates, benzodiazepines, or lithium within 14 days or 5 half-lives, whichever was longer, of randomization and at anytime throughout the study
* History of contraindications to anticholinergic agents (eg, bowel or urinary obstruction, stenosing peptic ulcers, narrow-angle glaucoma)
* History of allergy or intolerance to dibenzoxazepines (loxapine and amoxapine)
* History of extrapyramidal disorders, movement disorders including Parkinson's disease or neuroleptic malignant syndrome
* Female patients with a positive pregnancy test at screening or during randomization visit, or who were breastfeeding
* History within the past year of drug or alcohol dependence or abuse as defined by DSM IV
* History of syncope, unstable angina, myocardial infarction (within 6 months), congestive heart failure, or uncontrolled hypertension
* History of a major neurological disorder other than migraine (seizure disorder, subarachnoid bleeding, stroke, brain tumor, or transient ischemic attack)
* Any other disease(s), by history, physical examination, or laboratory abnormalities (including alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 2-fold the upper limit of normal, total bilirubin > 1.5 mg/dL, or creatinine > 1.8 mg/dL), that in the investigator's opinion, would present undue risk to the patient or could confound the interpretation of study results
* History of asthma or chronic obstructive lung disease or any use of an inhaler prescribed for wheezing or bronchospasm in the past 5 years
* Receipt of an investigational drug within 30 days prior to the screening visit
* Considered by the investigator, for any reason, to be an unsuitable candidate for receiving loxapine, or unable to use the inhalation device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K. Cady, MD, Principal Investigator — Clinvest; Peter J. Bellafiore, MD, Principal Investigator — CNS Research, Inc.; Arthur Elkind, MD, Principal Investigator — Elkind Headache Center
Locations (3):
- United States (3):
  - Roger K. Cady, Springfield, Missouri
  - Elkind Headache Center, Mount Vernon, New York
  - CNS Research, Inc., East Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inhaled Placebo | Inhaled Loxapine 1.25 mg | Inhaled Loxapine 2.5 mg
Started | 125 | 121 | 120
Completed | 125 | 121 | 120
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Placebo | Inhaled Loxapine 1.25 mg | Inhaled Loxapine 2.5 mg | Total
Number analyzed (Participants) | 125 | 121 | 120 | 366
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 125 | 121 | 120 | 366
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (12.14) | 41.2 (12.19) | 42 (12.74) | 41.5 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 100 | 41 | 229
  Male | 37 | 21 | 79 | 137
Region of Enrollment [Number; unit: participants]
  United States | 125 | 121 | 120 | 366

OUTCOME MEASURES:

1. Primary Outcome: Pain-Relief at 2 Hours Post-treatment
Description: Pain-Relief=pretreatment pain rating of 2 (moderate) or 3 (severe) and a rating of 0 (none) or 1 (mild) at the designated assessment time
Time Frame: 2 hours
Population: ITT with LOCF Population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Placebo | Inhaled Loxapine 1.25 mg | Inhaled Loxapine 2.5 mg
Number analyzed (Participants) | 124 | 121 | 119
Participants | 56 | 65 | 66

2. Secondary Outcome: Photophobia Free
Description: Free of Photophobia at 2 Hours Post-treatment
Time Frame: 2 hours
Population: ITT with LOCF Population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Placebo | Inhaled Loxapine 1.25 mg | Inhaled Loxapine 2.5 mg
Number analyzed (Participants) | 124 | 121 | 119
Participants | 59 | 47 | 54

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were considered treatment related from the first exposure to study treatment until 30 days after the last treatment
Description: Subjects were instructed to carry out self-assessment for adverse events from dosing through 24 hours and recored in the patient diary
Arm/Group | Inhaled Placebo | Inhaled Loxapine 1.25 mg | Inhaled Loxapine 2.5 mg
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/121 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/121 | 0/120
Other Adverse Events (participants affected / at risk) | 22/125 | 27/121 | 24/120
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Placebo (N=125) | Inhaled Loxapine 1.25 mg (N=121) | Inhaled Loxapine 2.5 mg (N=120)
Dysgeusia (Gastrointestinal disorders) | 6 (6) | 16 (16) | 10 (10)
Dizziness (Nervous system disorders) | 12 (12) | 8 (8) | 6 (6)
Somnolence (Nervous system disorders) | 4 (4) | 3 (3) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less